CLINICAL TRIAL: NCT02923791
Title: A Phase I, Randomized Open-label, 2-period, Parallel Arm Study To Assess The Immunogenicity Of Multiple Subcutaneous (SC) Doses Of "Filgrastim Hospira" (US) Or US-approved Neupogen(Registered) Reference Product In Healthy Volunteers
Brief Title: A Study in Healthy Volunteers to Assess Immune Response to Multiple Injections of Filgrastim Hospira or Neupogen Reference Product.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C1121012; FILGRASTIM IMMUNOGENICITY US (Other: Alias Study Number); COMPARATIVE IMMUNOGENICITY (Other: Alias Study Number)
Record Dates: First submitted 2016-09-30; First posted 2016-10-05 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Filgrastim Hospira (Experimental)
  Interventions: Biological: Filgrastim Hospira
- US-Approved Neupogen (Active Comparator)
  Interventions: Biological: US-Approved Neupogen

INTERVENTIONS:
Biological: Filgrastim Hospira — 5 consecutive daily doses (Days 1-5) in Period 1 and 1 dose (Day 1) in Period 2.
  Other Names: Filgrastim
  Arms: Filgrastim Hospira
Biological: US-Approved Neupogen — 5 consecutive daily doses (Days 1-5) in Period 1 and 1 dose (Day 1) in Period 2.
  Other Names: Filgrastim
  Arms: US-Approved Neupogen

SUMMARY:
This study compares the potential immunogenicity of two filgrastims, the proposed biosimilar Filgrastim Hospira (US) and the US-approved Neupogen reference product. Subjects will receive doses of one of the two filgrastims by injection of 5 micrograms/kilogram (mcg/kg). Subjects will receive 5 consecutive daily doses in Period 1 (Days 1-5) and a single dose on Day 1 of Period 2. Pre-dose and serial post-dose assessments of immunogenicity will be conducted each of the two study periods. In addition, safety assessments will be conducted throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
2. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Healthy male or female volunteers between 18 and 65 years of age (both inclusive).
4. Body mass index (BMI) between 19 and 30 kg/m2, inclusive, and body weight of not < 50 kg or >95 kg.
5. Subjects have abstained from the use of tobacco- or nicotine-containing products for at least 90 days prior to dosing and have a negative urine screen for cotinine at Screening.
6. Agrees to abstain from alcohol consumption for at least 48 hours prior to Day 1 of dosing in each study period and throughout the 5 days of study treatment and has a negative urine screen for alcohol at Screening.
7. Female subjects of non-childbearing potential must meet at least 1 of the following criteria:

   1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status will be confirmed by having a serum follicle-stimulating hormone (FSH) level confirming the postmenopausal state;
   2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
   3. Have medically confirmed ovarian failure. All other female subjects (including female subjects with tubal ligations) are considered to be of childbearing potential

Exclusion Criteria:

Subjects with any of the following characteristics/conditions will not be included in the study:

1. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
2. Participation in other studies involving an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product (whichever is longer) prior to study entry and/or during study participation.
3. Acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
4. Any active systemic or immunologic disease or condition, including but not limited to the following general categories: cardiovascular/pulmonary, hepatorenal, or systemic infection, or lactation.
5. History of malignancy or current malignancy with the exception of adequately treated squamous or basal cell carcinoma of the skin or cervical carcinoma in situ within 5 years.
6. Any disease or condition that might interfere with the absorption, distribution, metabolism, or excretion of the study drug or would place the subject at increased risk.
7. Hematologic laboratory abnormalities including leukocytosis (defined as total leukocytes >11,000/mcL), leukopenia (defined as total leukocytes <4000/mcL), or neutropenia (defined as absolute neutrophil count [ANC] <1500/mcL), or thrombocytopenia (defined as platelet count of <150/mcL).
8. Lacks adequate hepatic reserve as defined by aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≥ 1.5 x the upper limit of normal (ULN) of the reference lab; lack of renal reserve as defined by serum creatinine of ≥1.2 x ULN for reference lab or estimated glomerular filtration rate (eGFR) of ≤ 80 mg/min; or has known history of glomerulonephritis.
9. Clinically significant, as judged by the investigator, vital sign, or 12-lead electrocardiogram (ECG) abnormality.
10. History of biological growth factor exposure, including but not limited to filgrastim and other G-CSFs in the context of treatment, prophylaxis, peripheral blood stem cell mobilization, or previous investigational study setting.
11. Receipt of live vaccination, or exposure to communicable viral diseases such as chicken pox, varicella, or measles within the 4 weeks prior to Screening.
12. Surgery within the 4 months prior to Screening.
13. Use of any prescription medicine (with the exception of contraceptives) within 7 days or at least 5 half-lives, whichever is longer. Use of oral or parenteral anticoagulant or antiplatelet agents and corticosteroids should be specifically queried.
14. Administration of a drug by depot injection (with exception of depot contraception) within 30 days prior to the initial study drug administration or 5 half-lives of that drug, whichever is longer.
15. Use of over the counter medications, including aspirin and non-steroidal anti-inflammatory drugs, or natural preparations (dietary supplement or herbal product) within 7 days or at least 5 half-lives, whichever is longer. Vitamins and calcium supplements are allowed (not to exceed 100% daily value).
16. History of drug or alcohol abuse within 2 years prior to randomization, as determined by the investigator or a positive urine screen for drugs of abuse at Screening. Screening for drugs of abuse will minimally include cannabinoids, opiates, barbiturates, amphetamines, cocaine, and benzodiazepines.
17. Drug sensitivity, allergic reaction to, or known hypersensitivity/idiosyncratic reaction to E. coli-derived proteins, filgrastim, pegfilgrastim, other G-CSFs or any component of the product: subjects with the rare heredity problem of fructose intolerance are excluded due to the excipient sorbitol.
18. History of splenic rupture (or subject who is asplenic), pulmonary infiltrate or pneumonia, sickle cell disorders, chronic neutropenia, thrombocytopenia, or vasculitis.
19. Any clinically significant, as determined by the investigator, abnormal laboratory evaluations, including human immunodeficiency virus antibody (HIVAb), hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibody (HCVAb) and liver function taken at Screening. Negative HIVAb status will be confirmed at Screening and the results will be maintained confidentially by the study site.
20. Blood donation (including plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing OR had a transfusion of any blood product within 90 days prior to Screening.
21. Pregnant female subjects, breastfeeding female subjects, fertile male subjects and female subjects of childbearing potential who are unwilling or unable to use at least 1 highly effective method of contraception as outlined in the protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
22. Unwilling or unable to comply with the criteria in the Lifestyle Requirements section of the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2016-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with a negative baseline anti-drug antibody (ADA) test result and confirmed post-dose positive ADA test result at any time during the study. | 62 days (Period 1 Day 0 through Period 2 Day 31 or Final Visit)

SECONDARY OUTCOMES:
The proportion of subjects with a negative baseline ADA test result and post-dose positive neutralizing antibody result at any time during the study; | 62 days (Period 1 Day 0 through Period 2 Day 31 or Final Visit)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - SeaView Research, Inc., Coral Gables, Florida
  - Seaview Jacksonville LLC, Jacksonville, Florida
  - SeaView Research, Inc., Miami, Florida

REFERENCES:
- [Derived] Yao HM, Ottery FD, Borema T, Harris S, Levy J, May TB, Moosavi S, Zhang J, Summers M. PF-06881893 (Nivestym), a Filgrastim Biosimilar, Versus US-Licensed Filgrastim Reference Product (US-Neupogen(R)): Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Safety of Single or Multiple Subcutaneous Doses in Healthy Volunteers. BioDrugs. 2019 Apr;33(2):207-220. doi: 10.1007/s40259-019-00343-8. PMID 30900158
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C1121012&StudyName=A+Phase+I%2C+Randomized+Open-label%2C+2-period%2C+Parallel+Arm+Study+To+Assess+The+Immunogenicity+Of+Multiple+Subcutaneous+%28sc%29+Doses+Of+%E2%80%9Cfilgrastim+Hospira%E2%80%9D+%28us%29+Or+Us-approved+Neupogen%28registered%29+Reference+Product+In+Healthy+Volunteers